CLINICAL TRIAL: NCT04773613
Title: The Impact of Positioning on Bottle-feeding in Preterm Infants ≤34 Gestational Age. A Comparative Study of the Semi-elevated and Side-lying Position
Brief Title: The Impact of Positioning on Bottle-feeding in Preterm Infants. A Comparative Study PMMHHRI-2018/V/9-SZB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Anna Raczyńska, Principal Investigator, Polish Mother Memorial Hospital Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PMMHRI
Record Dates: First submitted 2021-01-30; First posted 2021-02-26 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-02

CONDITIONS: Bottle Feeding; Premature
Keywords: Premature Infant; Bottle Feeding; Side-lying Position; Semi-elevated Position; Oral Feeding
MeSH Terms: conditions — Bottle Feeding; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental SLP (Experimental): Infant placed in a SLP on the researcher's lap. Head of the infant symmetrically placed between the shoulders, supported by the researcher's. Shoulder girdle higher than the pelvic girdle, head and back in a straight line - a slight natural bend of the body is allowed. Legs bent at an angle of approx. 90° in the natural flexion of the knee and ankle joint. The infant's arms close to the midline (on the bottle or researcher's hands)
  Interventions: Other: Experimental SLP
- Experimental SEP (Other): Infant placed in a SEP on the researcher's lap. The head rests on the researcher's hand. Shoulder girdle higher than the pelvic girdle, head and back in a straight line at an angle of 30-45° to the ground - slight, natural body bend is allowed. Legs bent at an angle of approx. 90° in the natural flexion of the knee and ankle joint. The infant's arms close to the midline (on the bottle or researcher's hands)
  Interventions: Other: Experimental SEP

INTERVENTIONS:
Other: Experimental SLP — SLP was given to the infant during bottle-feeding.
  Arms: Experimental SLP
Other: Experimental SEP — SEP was given to the infant during bottle-feeding.
  Arms: Experimental SEP

SUMMARY:
One of the challenges of modern neonatology is to identify the right and effective method that can improve oral feeding. Optimal feeding position may contribute to improving the quality and safety of bottle-feeding in premature infants.

DETAILED DESCRIPTION:
PURPOSE: The aim of the study was to compare the advantages of semi-elevated (SEP) with side-lying positioning (SLP) during bottle-feeding of preterm infants.

METHOD: The study included forty two neonates (n=42) born ≤34 weeks of gestational age. Four bottle-feeding sessions were tested in each of the newborns: two in the SEP and two in the SLP. The position for the first study was randomly assigned, then positioning changed after each feeding session. In one day, only two consecutive feeding sessions which were included to the study in order to minimize fatigability as a disrupting factor. The levels of saturation (SpO2) and heart rate (HR) were measured as the parameters indicative of the newborn's physiological stability. The factors determining the qualitative aspect of feeding included the total time of declines of SpO2 ≤85%, level of the newborn's alertness according to the Neonatal Behavioral Assessment Scale (NBAS), and the occurrence of choking episodes. The proportion of milk consumed (volume of milk eaten relative to the expected volume) and the duration of the feeding and feeding session were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* circulatory and respiratory stability;
* readiness for oral feeding according to each child's Speech-Language Pathologist assessment;
* prematurely born infants who were in the process of being transferred from enteral nutrition (or enteral nutrition + parenteral nutrition) to full oral feeding and were fed orally at least 4- 6 times within twenty-four hours;
* parents gave informed consent to participate their infant in the study.

Exclusion Criteria:

* disorders which could significantly affect the feeding course, such as cleft lip and/or palate, facial paralysis and/or congenital defects of the facial skeleton;
* the presence of detected congenital abnormalities and metabolic diseases; low Apgar score (less than 5 points at the 5th and 10th minute of the measurement);
* administered analgesics, anticonvulsants and sedatives;
* <72 hours from extubation prior the trial;
* parents refusal to participate in the study or when bottle-feeding was not the parental preference.

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Physiological stability | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Oxygen saturation (SpO2) changes measured by using a pulse oximeter data
Physiological stability | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Heart rate (HR) changes measured by using a pulse oximeter data
Qualitative aspect of bottle-feeding | Measured during feeding
  Total time of declines of SpO2 ≤85%
Qualitative aspect of bottle-feeding | Measured 2 minutes before feeding session, in 3rd and 10th minutes of feeding, at the moment of finish of the feeding and in 10th minute after feeding (5 points of measurement)
  Level of the newborn's alertness changes according to the 6-point Neonatal Behavioral Assessment Scale, where individual points mean: 1 - quiet sleep, 2 - active sleep, 3 - drowsy, 4 - quiet alert, 5 - active alert, 6 - crying. This is descriptive, qualitative scale which shows changes of newborn's activity.
Qualitative aspect of bottle-feeding | Noticed during feeding
  Occurrence of choking episodes
Qualitative aspect of bottle-feeding | Measured from taking the baby out of bed before feeding to putting the baby to bed immediately after the intervention. Putting baby on parent's chest to kangaroo (Kangaroo Mother Care) after feeding instead to bed was also allowed.
  Duration of the feeding session
Qualitative aspect of bottle-feeding | Measured from insertion of the nipple to the infant's mouth to the moment when baby finish the feeding
  Duration of feeding
Qualitative aspect of bottle-feeding | Measured in 10th minute of feeding and on the finish of the feeding (2 points of measurement)
  Proportion of milk consumed (volume of milk eaten relative to the expected volume)

CONTACTS AND LOCATIONS:
Overall Officials: Anna D Raczyńska, MSc, Principal Investigator — Polish Mother's Memorial Hospital- Research Institute
Locations (1):
- Polish Mother's Memorial Hospital- Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT04773613/Prot_SAP_000.pdf